CLINICAL TRIAL: NCT06982742
Title: Development of a Mobile Health Application for Patients With Neuropathic Pain in Multiple Sclerosis and the Effect of the Application on Pain Intensity and Quality of Life
Brief Title: Effect of a Mobile Health App on Pain and Quality of Life in Patients With Neuropathic Pain in Multiple Sclerosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Meryem Kocaslan Toran (Other)
Collaborators: Uskudar University (Other); The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Sponsor-Investigator, Meryem Kocaslan Toran, Principal investigator, Uskudar University
Organization: Uskudar University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UskudarU-MS-PAINAPP-2025; TUBITAK 1002- 424S249 (Other Grant/Funding Number: TUBITAK)
Record Dates: First submitted 2025-05-13; First posted 2025-05-21 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; neuroparthic pain; quality opf life; mobile health aplication
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: Arm 1 Name: Mobile Health Application Group Intervention: Behavioral - Use of a Mobile Health Application Arm 2 Name: Standard Care Group Intervention: No Intervention - Standard Care
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 Name: Mobile Health Application Group (Intervention) (Experimental): Participants will use the mobile health application for 8 weeks.
  Interventions: Other: Mobile Health App for Neuropathic Pain Management in MS
- Arm 2 Name: Standard Care Group (Control) (No Intervention): Participants will receive standard care without the mobile health application.

INTERVENTIONS:
Other: Mobile Health App for Neuropathic Pain Management in MS — This intervention is a self-management mobile health application specifically designed for patients with Multiple Sclerosis who experience neuropathic pain. Unlike general symptom tracking apps, this application provides structured educational content on anti-inflammatory nutrition, physical activity, sleep hygiene, stress management, and smoking cessation. It includes goal-setting features, personalized reminders, symptom tracking tools, and feedback mechanisms to promote behavior change and self-efficacy. The intervention is designed based on Social Cognitive Theory, aiming to empower patients to actively manage their pain and improve their quality of life. T
  Arms: Arm 1 Name: Mobile Health Application Group (Intervention)

SUMMARY:
Multiple sclerosis (MS) is a chronic autoimmune disease affecting the central nervous system, leading to inflammation, neurodegeneration, and a range of physical and invisible symptoms. Among these, neuropathic pain significantly impairs quality of life but is often overlooked. Neuropathic pain in MS is associated with increased central sensitivity, neuroinflammation, and lifestyle factors such as unhealthy diet, physical inactivity, poor sleep, stress, and smoking. While pharmacological treatments are commonly used, they often provide limited long-term relief and may carry risks such as dependence and side effects.

Growing evidence highlights the importance of non-pharmacological, self-management interventions that promote lifestyle changes. Digital health technologies, particularly mobile health (mHealth) applications, have emerged as accessible tools to support self-management, allowing individuals to take an active role in managing their symptoms and improving their well-being. However, existing mHealth applications often lack scientifically validated content, do not specifically address neuropathic pain, and have limited user-centered design features.

This study aims to develop a self-management-based mHealth application tailored for patients with MS experiencing neuropathic pain. Grounded in Bandura's Social Cognitive Theory, the application will provide educational content, symptom tracking, goal-setting tools, and behavior change strategies covering topics such as nutrition, physical activity, sleep hygiene, stress management, and smoking cessation. The application seeks to improve self-efficacy, reduce pain intensity, and enhance quality of life.

The study will be conducted as a randomized controlled trial. Participants will be randomly assigned to an intervention group (using the mHealth application for eight weeks) or a control group (receiving standard care). Primary outcomes include changes in pain intensity and quality of life. The study hypothesizes that using the mobile application will reduce pain intensity and improve quality of life compared to standard care.

Additionally, the study sets measurable success criteria for the development and evaluation of the application, including expert and user evaluations of content quality, usability, and user satisfaction. The findings aim to contribute to the literature on integrative pain management and demonstrate the

DETAILED DESCRIPTION:
This randomized controlled trial aims to evaluate the efficacy of a self-management-based mobile health application designed for individuals with Multiple Sclerosis (MS) who experience neuropathic pain. Neuropathic pain, affecting up to 58% of MS patients, is associated with neuroinflammation, central sensitization, and oxidative stress, often exacerbated by lifestyle factors such as poor diet, inactivity, poor sleep hygiene, stress, and smoking.

The proposed mobile application is built upon Bandura's Social Cognitive Theory and includes five core modules: self-monitoring, health education, goal-setting, skill-building, and professional support access. The app supports behavior change and provides targeted education on anti-inflammatory nutrition, physical activity, sleep hygiene, stress management, and smoking cessation, aiming to reduce neuropathic pain intensity and improve quality of life.

The app is developed using Flutter/Dart and includes interactive features such as pain diaries, daily goals, reminders, and feedback mechanisms. Educational materials are prepared with input from an interdisciplinary expert panel and validated using DISCERN and HEMDA tools.

The intervention phase will last eight weeks. Patients will be randomized into either the intervention group (app users) or the control group (usual care). Primary outcomes include reduction in pain intensity (VAS) and improvement in quality of life (MSQOL-54). Secondary measures include changes in depression (BDI), insomnia (ISI), fatigue (FSS), and self-management (MSSM).

This project addresses an unmet need for digital, non-pharmacological, evidence-based strategies to support MS patients with neuropathic pain and aims to offer a scalable and accessible solution for long-term self-management.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years of age or older,
* Having a definitive diagnosis of MS according to the McDonald 2017 criteria,
* Owning a smartphone with an Android operating system,
* Having an Expanded Disability Status Scale (EDSS) score ≤ 5*,
* Being able to communicate in Turkish,
* Being literate,
* No neurological symptoms that could impair smartphone use (e.g., tremor),
* Pain Detect Pain Questionnaire score of 19 or higher,
* Neuropathic Pain Questionnaire score of 4 or higher,
* Beck Depression Scale score below 17, *EDSS scores determined by a physician's evaluation will be considered.

Exclusion Criteria:

* Having undergone surgical interventions on the musculoskeletal system (for at least six months),
* Having a known neurological disorder (epilepsy, dementia)*,
* Having vision or hearing problems that could affect test performance*,
* Chronic pain not attributable to neuropathic causes (cancer, carpal tunnel syndrome, postherpetic neuralgia)*,
* Peripheral vascular complications due to diabetes or other etiologies*,
* Participation in supervised exercise, home exercise, group exercise, etc., as part of physical therapy*,
* Participation in psychological therapies (cognitive and/or behavioral therapy, biofeedback), *
* Participation in mind-body practices (yoga, tai chi, etc.),*
* Participation in acupuncture, *
* Receiving invasive treatments (e.g., injections, nerve blocks, spinal cord stimulators, parenteral medications, etc.) *, * Patient self-report and medical records will be used as the basis for inclusion; patients with observed vision or hearing impairments during testing will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Reduction in Neuropathic Pain Intensity Measured by Visual Analog Scale (VAS) | Baseline and 8 weeks after intervention start
  Assessment of change in neuropathic pain intensity using the Visual Analog Scale (VAS), scored from 0 (no pain) to 10 (worst imaginable pain), comparing baseline and 8-week follow-up scores between the intervention and control groups in a randomized controlled trial.

SECONDARY OUTCOMES:
Improvement in Quality of Life Measured by Multiple Sclerosis Quality of Life-54 (MSQOL-54) | Baseline and 8 weeks after intervention start
  Assessment of change in health-related quality of life using the MSQOL-54 scale, comparing baseline and 8-week follow-up scores between the intervention and control groups in a randomized controlled trial.

CONTACTS AND LOCATIONS:
Locations (1):
- Uskudar University, Faculty of Health Sciences, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No